CLINICAL TRIAL: NCT05010330
Title: Multi-omics Combined With Clinical Data Analysis to Identify Prognostic Biomarkers of Lung Cancer
Brief Title: Identify Prognostic Biomarkers of Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MKM2021-720
Record Dates: First submitted 2021-07-27; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer; Lung Adenocarcinoma; Lung Squamous Cell Carcinoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — In this study ,we planned to collect plasm from the two cohorts, and lung cancer tissues and para-carcinoma tissue from lung cancer patients who had a tumor excision
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy control: healthy people
- lung cancer: patients diagnosed with lung cancer

SUMMARY:
Multi-omics and Clinical Data Analysis is potential to predict the prognosis of lung cancer patients.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death in China. In order to improve prognosis of lung cancer as well as provide new therapeutic targets, the identification of effective biomarkers for the prognosis of lung cancer is of great significance. It has been reported that some small molecules such as lncRNA, circRNA and polypeptides in human plasm have good prospects in diagnosing or evaluating the stage of diseases. In this study, we planned to use multi-omics combined with clinical data to discovery some small molecules that are potential to predict the prognosis of lung cancer patients. In addition, we want to construct a new risk score model that provide a candidate model for prognostic evaluation of lung cancer. And we hope our study can provide insights for precision immunotherapy of lung cancer by exploring the differences in clinical characteristics, tumor mutation burden, and tumor immune cell infiltration between different risk score groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer;
* Untreated lung cancer patients;
* No history of chronic or serious diseases, such as cardiovascular disease, liver disease, kidney disease, respiratory disease, blood disease, lymphatic disease, endocrine disease, immune disease, mental disease, neuromuscular disease, gastrointestinal system disease, etc.

Exclusion Criteria:

* Patients with other tumors;
* Lung cancer patients who had been treated;
* Abnormal liver and kidney function;
* Acute and chronic infectious diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged between 18 and 80 years old. Patients with diagnosis of lung cancer or healthy controls without any history of tumor will be eligible for our enrollment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Identify some prognostic biomarkers in lung cancer. | 1 week
  1. Our study will identify some biomarkers that can predict the prognosis of lung cancer patients.
  2. Our study will construct a new risk score model that provide a candidate model for prognostic evaluation of lung cancer.
  3. Our research will provide insights for precision immunotherapy of lung cancer by exploring the differences in clinical characteristics, tumor mutation burden, and tumor immune cell infiltration between different risk score groups.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Huang, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University school of medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Zhang Y, Yang M, Ng DM, Haleem M, Yi T, Hu S, Zhu H, Zhao G, Liao Q. Multi-omics Data Analyses Construct TME and Identify the Immune-Related Prognosis Signatures in Human LUAD. Mol Ther Nucleic Acids. 2020 Sep 4;21:860-873. doi: 10.1016/j.omtn.2020.07.024. Epub 2020 Jul 23. PMID 32805489